CLINICAL TRIAL: NCT02529527
Title: MyFamilyPlan: A Patient-Centered Web-based Preconception Health Education Tool
Brief Title: Web-based Preconception Health Education Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB#15-001313
Record Dates: First submitted 2015-05-19; First posted 2015-08-20 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Reproductive Health

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- MyFamilyPlan (Experimental): Web-based health education tool (interactive self-assessment) provided for participant completion 7-10 days prior to a scheduled primary care visit.
  Interventions: Behavioral: MyFamilyPlan
- Control (No Intervention): Standard preconception health education document provided for participant review 7-10 days prior to a scheduled primary care visit.

INTERVENTIONS:
Behavioral: MyFamilyPlan — Web-based preconception health education tool (interactive self-assessment) - to be completed by patient
  Arms: MyFamilyPlan

SUMMARY:
Strong evidence supports that preconception care, or care to optimize a woman's health health prior to pregnancy, can improve birth outcomes. Preconception health counseling covers a broad range of topics, including: desire for pregnancy, obstetric history, nutrition, vaccinations, sexual health, chronic disease, substance abuse, mental health and contraception. Despite calls from public health organizations and experts in the field for universal access to preconception care, most US women do not receive any health counseling to prepare for pregnancy. Given that approximately half of US pregnancies are unintended, it is critical that routine primary care serve as a venue for the provision of this important service. From a patient's perspective, improving preconception health involves many health behavior changes. As such, patient engagement and education regarding preconception health must be a primary focus. Several preconception health promotion tools have been developed for patients to date; few are truly patient-centered and even fewer have been rigorously evaluated.

This study presents MyFamilyPlan - a novel, web-based, patient centered preconception health education tool designed for women of reproductive age receiving primary care. MyFamilyPlan is truly innovative in two key ways:

* MyFamilyPlan is a web-based preconception health self-assessment. This will allow for the employment of skip logic to individualize the questionnaire and subsequent health recommendations for each patient.
* Recognizing that preconception care is relevant to all women "at risk" of pregnancy, MyFamilyPlan has been designed for utilization in a primary care setting.

This preconception health education tool will be tested using a randomized controlled design. This study will measure whether or not exposure to MyFamilyPlan promotes the discussion of preconception health issues in primary care encounters (primary outcome). It will also evaluate whether the intervention affects participant self-efficacy in planning a healthy pregnancy, and relevant health behaviors (secondary outcome). The study proposed here will improve the quality of evidence for preconception health education tools. Should it demonstrate effectiveness, it will also result in a new tool that could be made more widely available to promote preconception health.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years of age
* English-speaking
* Non-pregnant
* Capable of pregnancy (i.e., no previous hysterectomy or sterilization procedure)
* Scheduled primary care visit in health system in the upcoming 7-10 days
* Active email address

Exclusion Criteria;

* Currently pregnant

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 292 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Proportion of women (intervention vs. control) reporting discussion of preconception health with provider at the primary care visit | 7-10 days after exposure to intervention
  Patient-reported discussion of preconception health with a provider at the primary care visit (measured by post-intervention patient survey: yes/no item)

SECONDARY OUTCOMES:
Numerical change in reported patient self-efficacy with respect to pregnancy planning before and after exposure to education tool (score range: 0-60) | 7-10 days after exposure to intervention
  Change in self-efficacy score (patient-rated) after exposure to intervention or control (measured by change in 6-item validated Reproductive Health and Behaviors self-efficacy score between pre-intervention patient survey and post-intervention patient survey)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Derived] Batra P, Mangione CM, Cheng E, Steers WN, Nguyen TA, Bell D, Kuo AA, Gregory KD. A Cluster Randomized Controlled Trial of the MyFamilyPlan Online Preconception Health Education Tool. Am J Health Promot. 2018 May;32(4):897-905. doi: 10.1177/0890117117700585. Epub 2017 Apr 10. PMID 28391703